CLINICAL TRIAL: NCT00778492
Title: Thrombelastogram and Predicting Microvascular Bleeding in Patients Receiving Antiplatelet Medication Undergoing Cardiac Surgery
Brief Title: Thrombelastogram in Patients Receiving Antiplatelet Medication Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sergey Preisman, MD, Sheba Medical Center
Other Study IDs: SHEBA-08-5119-SP-CTIL
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Bleeding
Keywords: Thrombelastogram; Microvascular bleeding; antiplatelet medication; cardiac surgery; consumption of blood products; preoperative platelet mapping derived from modified TEG; postoperative bleeding
MeSH Terms: conditions — Hemorrhage; Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment: Patients with the history of ingestion of aspirin and/or ADP receptor antagonist (clopidogrel or ticlopidine) for at least 7 days prior the surgery. All patients undergoing cardiac surgery with the use of cardiopulmonary bypass on elective and urgent basis.

SUMMARY:
Study Objective is to correlate the results of preoperative platelet mapping derived from modified TEG with clinically significant postoperative bleeding and consumption of blood products.

DETAILED DESCRIPTION:
Study Design:

Prospective observational study with blinded assessment of study endpoint variables. Collection of information concerning study endpoints will be performed by the investigator blinded to the results of preoperative testing of platelet function. The information will be collected from 60 patients undergoing cardiac surgery in the Department of Cardiac Surgery of Sheba Medical Center.

Study endpoints

1. Primary endpoint- resternotomy for bleeding after the surgery.
2. Secondary endpoints- chest tube output during first 24 hours after the surgery; consumption of blood products during first 3 postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery with the history of aspirin and/or ADP receptor antagonist for at least 7 days prior the surgery

Exclusion Criteria:

* Emergent surgery
* Heart transplant surgery
* Implantation of ventricular assist devices
* Enrollment into conflicting study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the history of ingestion of aspirin and/or ADP receptor antagonist (clopidogrel or ticlopidine) for at least 7 days prior the surgery. All patients undergoing cardiac surgery with the use of cardiopulmonary bypass on elective and urgent basis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-10 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Re-sternotomy d/t Bleeding | Hospitalization Period

SECONDARY OUTCOMES:
Chest tube output during first 24 hours after the surgery | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Preisman, MD, Principal Investigator — Sheba Medical Center; Alexander Kogan, MD, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel